CLINICAL TRIAL: NCT00673816
Title: Pilot Study of Sunitinib Malate for Advanced Ocular Disease of Von Hippel-Lindau Syndrome
Brief Title: Sunitinib Malate to Treat Advanced Eye Disease in Patients With Von Hippel-Lindau Syndrome
Acronym: VHL3
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inability to recruit and adequate number of participants
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080129; 08-EI-0129 (Other: National Eye Institute)
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2011-11

CONDITIONS: Von Hippel-Lindau Syndrome
Keywords: Von Hippel Lindau; Sunitinib Malate; Sutent; Von Hippel-Lindau Syndrome; VHL
MeSH Terms: conditions — von Hippel-Lindau Disease | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib Malate (Experimental): Participants were expected to receive 9 months of sunitinib malate therapy administered in 6 cycles. Each cycle consisted of a daily oral dose of 50 mg sunitinib malate for 4 weeks followed by a 2-week rest period).
  Interventions: Drug: Sunitinib Malate

INTERVENTIONS:
Drug: Sunitinib Malate — Participants were expected to receive 9 months of sunitinib malate therapy administered in 6 cycles. Each cycle consisted of a daily oral dose of 50 mg sunitinib malate for 4 weeks followed by a 2-week rest period).

SUMMARY:
This open-label study will pilot the use of systemic sunitinib malate, a dual inhibitor of vascular endothelial growth factor (VEGF) and platelet derived growth factor (PDGF), in five participants with Von Hippel-Lindau (VHL) to investigate its potential efficacy as a treatment for retinal angiomas. Participants will have visual dysfunction with either visual acuity loss or visual field loss from retinal angiomas secondary to genetically confirmed VHL. This open-label study will pilot the use of systemic sunitinib malate in five participants to investigate its potential efficacy as a treatment for retinal angiomas associated with VHL. Participants will receive nine months of sunitinib malate therapy (six cycles total - one cycle consists of 50 mg oral dose once daily for four weeks followed by a two week rest period). The primary outcome will be a change in the best-corrected visual acuity of more than or equal to 15 letters from baseline to the Week 36 visit. The secondary ocular outcomes will focus on retinal thickness and leakage of the retinal angioma at the Week 36 visit. Optical coherence tomography will document changes in retinal thickening and fluorescein angiography will be used to determine leakage of the retinal angioma.

ELIGIBILITY:
Inclusion Criteria

1. Participant must understand and sign the informed consent.
2. Participant must be at least 18 years of age.
3. Participant must have genetically confirmed VHL disease.
4. Participant must have an optic nerve angioma secondary to VHL in one or both eyes.
5. Participant must have an optic nerve tumor that has caused any visual field depression on microperimetry-1 that correlates with the retinal angioma OR the participant clinically may have hard exudates correlating with the retinal angioma OR has best-corrected visual acuity of 20/40 or worse in the study eye.
6. Participant must have clear ocular media and adequate pupillary dilation to permit good quality stereoscopic fundus photography.
7. All women of childbearing potential must have a negative urine pregnancy test at baseline, and have regular negative pregnancy testing while taking sunitinib malate. (Sunitinib malate has the potential for teratogenic or abortifacient effects, and no data regarding its safety in pregnant women are available).
8. All women of childbearing potential who are sexually active and all men who are sexually active are required to use two forms of birth control during the course of the study.
9. Participants must have normal organ and marrow function as defined below: WBC count ≥ 3,000/µL, absolute neutrophil count ≥ 1,500/µL, platelet count ≥ 100,000/µL, HGB> 10g/dl, serum creatinine ≤ 2.0 or measured 24 hr. creatinine clearance > 50 ml/min, AST and ALT < 2.5 x ULN, total bilirubin ≤ ULN (< 3 x NL in participants with Gilbert's disease).
10. Participant must have a negative HbsAg and nonreactive HCV.
11. Participant must have a negative HIV-1, as potential pharmacokinetic interactions of drugs used to treat HIV, such as anti-retroviral drugs, with sunitinib malate are unknown.
12. Participant must be at least four weeks from completion of any investigational therapy for VHL.
13. Participant must have an ECOG performance score of 0-2. (See Appendix 3 - ECOG Performance Criteria).
14. Participant has recovered from the acute toxicities of prior treatment for VHL.

Exclusion Criteria

1. Participant has a history (within past five years) or evidence of severe cardiac disease including heart failure that meets New York Heart Association (NYHA) class III and IV definitions, uncontrolled dysrhythmias, dysrhythmias requiring anti-arhythmic drugs or has active ischemic heart disease including myocardial infarction and poorly controlled angina within 12 months of study entry.
2. Participant has a history of serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation, ≥ three beats in a row) or left ventricular ejection fraction ≤ 40%.
3. Participant has a history of serious intercurrent medical illness.
4. Participant had transient ischemic attacks or cerebrovascular accident within 12 months of study entry.
5. Participant has hypertension that cannot be controlled with medications (persistent elevation of systolic BP > 150 or diastolic BP > 100 mmHg despite optimal medical therapy).
6. Participant is on therapeutic anticoagulation, including aspirin.
7. Participant who is breast-feeding, as there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sunitinib malate.
8. Participant has received any major surgical procedures within one month of study entry or has surgical scars that have not healed.
9. Participant has a known serious allergy to fluorescein dye.
10. Participant is currently taking drugs or ingesting food that affect sunitinib malate plasma concentrations: strong inhibitors of the CYP3A4 family (e.g., ketoconazole, itraconazole, clarithromycin, atazanavir, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, grapefruit juice) and/or inducers of the CYP3A4 family (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, St. John's Wort).
11. Participant has had a prior or concomitant non-VHL-associated malignancy with the exception of adequately treated basal or squamous cell carcinoma of the skin or any other malignancy from which the patient has remained disease free for more than five years.
12. Participant has had chemotherapy or radiotherapy within four weeks (six weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (to Grade 1 or less toxicity according to CTCAE 3.0) due to agents administered more than four weeks earlier.
13. Participant is receiving other investigational agents.
14. Participants with known brain metastases (except when adequately controlled, i.e., have not grown in size, for ≥ 6 months before enrollment), not including hemangioblastoma, a known VHL complication of the brain.
15. Participant has a known bleeding disorder.
16. Participant is currently taking sunitinib malate or has taken sunitinib malate in the past.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Meyerle, MD, Principal Investigator — NEI/NIH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Siemeister G, Weindel K, Mohrs K, Barleon B, Martiny-Baron G, Marme D. Reversion of deregulated expression of vascular endothelial growth factor in human renal carcinoma cells by von Hippel-Lindau tumor suppressor protein. Cancer Res. 1996 May 15;56(10):2299-301. PMID 8625303
- [Background] Iliopoulos O, Levy AP, Jiang C, Kaelin WG Jr, Goldberg MA. Negative regulation of hypoxia-inducible genes by the von Hippel-Lindau protein. Proc Natl Acad Sci U S A. 1996 Oct 1;93(20):10595-9. doi: 10.1073/pnas.93.20.10595. PMID 8855223
- [Background] Gnarra JR, Zhou S, Merrill MJ, Wagner JR, Krumm A, Papavassiliou E, Oldfield EH, Klausner RD, Linehan WM. Post-transcriptional regulation of vascular endothelial growth factor mRNA by the product of the VHL tumor suppressor gene. Proc Natl Acad Sci U S A. 1996 Oct 1;93(20):10589-94. doi: 10.1073/pnas.93.20.10589. PMID 8855222
- [Background] Dahr SS, Cusick M, Rodriguez-Coleman H, Srivastava SK, Thompson DJ, Linehan WM, Ferris FL 3rd, Chew EY. Intravitreal anti-vascular endothelial growth factor therapy with pegaptanib for advanced von Hippel-Lindau disease of the retina. Retina. 2007 Feb;27(2):150-8. doi: 10.1097/IAE.0b013e318030a290. PMID 17290195
- [Background] Kurban G, Hudon V, Duplan E, Ohh M, Pause A. Characterization of a von Hippel Lindau pathway involved in extracellular matrix remodeling, cell invasion, and angiogenesis. Cancer Res. 2006 Feb 1;66(3):1313-9. doi: 10.1158/0008-5472.CAN-05-2560. PMID 16452184
- [Background] Aiello LP, George DJ, Cahill MT, Wong JS, Cavallerano J, Hannah AL, Kaelin WG Jr. Rapid and durable recovery of visual function in a patient with von hippel-lindau syndrome after systemic therapy with vascular endothelial growth factor receptor inhibitor su5416. Ophthalmology. 2002 Sep;109(9):1745-51. doi: 10.1016/s0161-6420(02)01159-4. PMID 12208726
- [Background] Girmens JF, Erginay A, Massin P, Scigalla P, Gaudric A, Richard S. Treatment of von Hippel-Lindau retinal hemangioblastoma by the vascular endothelial growth factor receptor inhibitor SU5416 is more effective for associated macular edema than for hemangioblastomas. Am J Ophthalmol. 2003 Jul;136(1):194-6. doi: 10.1016/s0002-9394(03)00101-6. PMID 12834696
- [Background] Seizinger BR, Rouleau GA, Ozelius LJ, Lane AH, Farmer GE, Lamiell JM, Haines J, Yuen JW, Collins D, Majoor-Krakauer D, et al. Von Hippel-Lindau disease maps to the region of chromosome 3 associated with renal cell carcinoma. Nature. 1988 Mar 17;332(6161):268-9. doi: 10.1038/332268a0. PMID 2894613
- [Background] Maher ER, Bentley E, Yates JR, Latif F, Lerman M, Zbar B, Affara NA, Ferguson-Smith MA. Mapping of the von Hippel-Lindau disease locus to a small region of chromosome 3p by genetic linkage analysis. Genomics. 1991 Aug;10(4):957-60. doi: 10.1016/0888-7543(91)90185-h. PMID 1680799
- [Background] MELMON KL, ROSEN SW. LINDAU'S DISEASE. REVIEW OF THE LITERATURE AND STUDY OF A LARGE KINDRED. Am J Med. 1964 Apr;36:595-617. doi: 10.1016/0002-9343(64)90107-x. No abstract available. PMID 14142412
- [Background] Horton WA, Wong V, Eldridge R. Von Hippel-Lindau disease: clinical and pathological manifestations in nine families with 50 affected members. Arch Intern Med. 1976 Jul;136(7):769-77. doi: 10.1001/archinte.136.7.769. PMID 945722
- [Background] Hardwig P, Robertson DM. von Hippel-Lindau disease: a familial, often lethal, multi-system phakomatosis. Ophthalmology. 1984 Mar;91(3):263-70. doi: 10.1016/s0161-6420(84)34304-4. PMID 6538954
- [Background] Green JS, Bowmer MI, Johnson GJ. Von Hippel-Lindau disease in a Newfoundland kindred. CMAJ. 1986 Jan 15;134(2):133-8, 146. PMID 3942913
- [Background] Ridley M, Green J, Johnson G. Retinal angiomatosis: the ocular manifestations of von Hippel-Lindau disease. Can J Ophthalmol. 1986 Dec;21(7):276-83. PMID 3801976
- [Background] Lamiell JM, Salazar FG, Hsia YE. von Hippel-Lindau disease affecting 43 members of a single kindred. Medicine (Baltimore). 1989 Jan;68(1):1-29. doi: 10.1097/00005792-198901000-00001. PMID 2642584
- [Background] Maher ER, Yates JR, Harries R, Benjamin C, Harris R, Moore AT, Ferguson-Smith MA. Clinical features and natural history of von Hippel-Lindau disease. Q J Med. 1990 Nov;77(283):1151-63. doi: 10.1093/qjmed/77.2.1151. PMID 2274658
- [Background] McDonald HR, Schatz H, Johnson RN, Abrams GW, Brown GC, Brucker AJ, Han DP, Lewis H, Mieler WF, Meyers S. Vitrectomy in eyes with peripheral retinal angioma associated with traction macular detachment. Ophthalmology. 1996 Feb;103(2):329-35 ; discussion 334-5. doi: 10.1016/s0161-6420(96)30696-9. PMID 8594522
- [Background] Kaelin WG Jr. Molecular basis of the VHL hereditary cancer syndrome. Nat Rev Cancer. 2002 Sep;2(9):673-82. doi: 10.1038/nrc885. PMID 12209156
- [Background] Rosenblatt MI, Azar DT. Anti-angiogenic therapy: Prospects for treatment of ocular tumors. Semin Ophthalmol. 2006 Jul-Sep;21(3):151-60. doi: 10.1080/08820530500350787. PMID 16912013
- [Background] Alvarez RH, Kantarjian HM, Cortes JE. Biology of platelet-derived growth factor and its involvement in disease. Mayo Clin Proc. 2006 Sep;81(9):1241-57. doi: 10.4065/81.9.1241. PMID 16970222
- [Background] Guo P, Hu B, Gu W, Xu L, Wang D, Huang HJ, Cavenee WK, Cheng SY. Platelet-derived growth factor-B enhances glioma angiogenesis by stimulating vascular endothelial growth factor expression in tumor endothelia and by promoting pericyte recruitment. Am J Pathol. 2003 Apr;162(4):1083-93. doi: 10.1016/S0002-9440(10)63905-3. PMID 12651601
- [Background] Morabito A, De Maio E, Di Maio M, Normanno N, Perrone F. Tyrosine kinase inhibitors of vascular endothelial growth factor receptors in clinical trials: current status and future directions. Oncologist. 2006 Jul-Aug;11(7):753-64. doi: 10.1634/theoncologist.11-7-753. PMID 16880234
- [Background] Mendel DB, Laird AD, Xin X, Louie SG, Christensen JG, Li G, Schreck RE, Abrams TJ, Ngai TJ, Lee LB, Murray LJ, Carver J, Chan E, Moss KG, Haznedar JO, Sukbuntherng J, Blake RA, Sun L, Tang C, Miller T, Shirazian S, McMahon G, Cherrington JM. In vivo antitumor activity of SU11248, a novel tyrosine kinase inhibitor targeting vascular endothelial growth factor and platelet-derived growth factor receptors: determination of a pharmacokinetic/pharmacodynamic relationship. Clin Cancer Res. 2003 Jan;9(1):327-37. PMID 12538485
- [Background] Motzer RJ, Michaelson MD, Redman BG, Hudes GR, Wilding G, Figlin RA, Ginsberg MS, Kim ST, Baum CM, DePrimo SE, Li JZ, Bello CL, Theuer CP, George DJ, Rini BI. Activity of SU11248, a multitargeted inhibitor of vascular endothelial growth factor receptor and platelet-derived growth factor receptor, in patients with metastatic renal cell carcinoma. J Clin Oncol. 2006 Jan 1;24(1):16-24. doi: 10.1200/JCO.2005.02.2574. Epub 2005 Dec 5. PMID 16330672
- [Background] O'Farrell AM, Foran JM, Fiedler W, Serve H, Paquette RL, Cooper MA, Yuen HA, Louie SG, Kim H, Nicholas S, Heinrich MC, Berdel WE, Bello C, Jacobs M, Scigalla P, Manning WC, Kelsey S, Cherrington JM. An innovative phase I clinical study demonstrates inhibition of FLT3 phosphorylation by SU11248 in acute myeloid leukemia patients. Clin Cancer Res. 2003 Nov 15;9(15):5465-76. PMID 14654525
- [Background] Abrams TJ, Murray LJ, Pesenti E, Holway VW, Colombo T, Lee LB, Cherrington JM, Pryer NK. Preclinical evaluation of the tyrosine kinase inhibitor SU11248 as a single agent and in combination with "standard of care" therapeutic agents for the treatment of breast cancer. Mol Cancer Ther. 2003 Oct;2(10):1011-21. PMID 14578466
- [Background] Murray LJ, Abrams TJ, Long KR, Ngai TJ, Olson LM, Hong W, Keast PK, Brassard JA, O'Farrell AM, Cherrington JM, Pryer NK. SU11248 inhibits tumor growth and CSF-1R-dependent osteolysis in an experimental breast cancer bone metastasis model. Clin Exp Metastasis. 2003;20(8):757-66. doi: 10.1023/b:clin.0000006873.65590.68. PMID 14713109
- [Background] Sakamoto KM. Su-11248 Sugen. Curr Opin Investig Drugs. 2004 Dec;5(12):1329-39. PMID 15648955
- [Background] Abrams TJ, Lee LB, Murray LJ, Pryer NK, Cherrington JM. SU11248 inhibits KIT and platelet-derived growth factor receptor beta in preclinical models of human small cell lung cancer. Mol Cancer Ther. 2003 May;2(5):471-8. PMID 12748309
- [Background] Schueneman AJ, Himmelfarb E, Geng L, Tan J, Donnelly E, Mendel D, McMahon G, Hallahan DE. SU11248 maintenance therapy prevents tumor regrowth after fractionated irradiation of murine tumor models. Cancer Res. 2003 Jul 15;63(14):4009-16. PMID 12873999
- [Background] Faivre S, Delbaldo C, Vera K, Robert C, Lozahic S, Lassau N, Bello C, Deprimo S, Brega N, Massimini G, Armand JP, Scigalla P, Raymond E. Safety, pharmacokinetic, and antitumor activity of SU11248, a novel oral multitarget tyrosine kinase inhibitor, in patients with cancer. J Clin Oncol. 2006 Jan 1;24(1):25-35. doi: 10.1200/JCO.2005.02.2194. Epub 2005 Nov 28. PMID 16314617
- [Background] Motzer RJ, Rini BI, Bukowski RM, Curti BD, George DJ, Hudes GR, Redman BG, Margolin KA, Merchan JR, Wilding G, Ginsberg MS, Bacik J, Kim ST, Baum CM, Michaelson MD. Sunitinib in patients with metastatic renal cell carcinoma. JAMA. 2006 Jun 7;295(21):2516-24. doi: 10.1001/jama.295.21.2516. PMID 16757724
- [Background] Bello CL, Sherman L, Zhou J, Verkh L, Smeraglia J, Mount J, Klamerus KJ. Effect of food on the pharmacokinetics of sunitinib malate (SU11248), a multi-targeted receptor tyrosine kinase inhibitor: results from a phase I study in healthy subjects. Anticancer Drugs. 2006 Mar;17(3):353-8. doi: 10.1097/00001813-200603000-00015. PMID 16520665
- [Background] Motzer RJ, Hoosen S, Bello CL, Christensen JG. Sunitinib malate for the treatment of solid tumours: a review of current clinical data. Expert Opin Investig Drugs. 2006 May;15(5):553-61. doi: 10.1517/13543784.15.5.553. PMID 16634693
- [Background] Escudier B, Chevreau C, Lasset C, Douillard JY, Ravaud A, Fabbro M, Caty A, Rossi JF, Viens P, Bergerat JP, Savary J, Negrier S. Cytokines in metastatic renal cell carcinoma: is it useful to switch to interleukin-2 or interferon after failure of a first treatment? Groupe Francais d'Immunotherape. J Clin Oncol. 1999 Jul;17(7):2039-43. doi: 10.1200/JCO.1999.17.7.2039. PMID 10561255
- [Background] Motzer RJ, Hutson TE, Tomczak P, Michaelson MD, Bukowski RM, Rixe O, Oudard S, Negrier S, Szczylik C, Kim ST, Chen I, Bycott PW, Baum CM, Figlin RA. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma. N Engl J Med. 2007 Jan 11;356(2):115-24. doi: 10.1056/NEJMoa065044. PMID 17215529
- [Background] Corless CL, McGreevey L, Town A, Schroeder A, Bainbridge T, Harrell P, Fletcher JA, Heinrich MC. KIT gene deletions at the intron 10-exon 11 boundary in GI stromal tumors. J Mol Diagn. 2004 Nov;6(4):366-70. doi: 10.1016/S1525-1578(10)60533-8. PMID 15507676
- [Background] Heinrich MC, Corless CL, Demetri GD, Blanke CD, von Mehren M, Joensuu H, McGreevey LS, Chen CJ, Van den Abbeele AD, Druker BJ, Kiese B, Eisenberg B, Roberts PJ, Singer S, Fletcher CD, Silberman S, Dimitrijevic S, Fletcher JA. Kinase mutations and imatinib response in patients with metastatic gastrointestinal stromal tumor. J Clin Oncol. 2003 Dec 1;21(23):4342-9. doi: 10.1200/JCO.2003.04.190. PMID 14645423
- [Background] Blanke CD, Corless CL. State-of-the art therapy for gastrointestinal stromal tumors. Cancer Invest. 2005;23(3):274-80. doi: 10.1081/cnv-200055972. PMID 15945512
- [Background] Van Glabbeke M, Verweij J, Casali PG, Le Cesne A, Hohenberger P, Ray-Coquard I, Schlemmer M, van Oosterom AT, Goldstein D, Sciot R, Hogendoorn PC, Brown M, Bertulli R, Judson IR. Initial and late resistance to imatinib in advanced gastrointestinal stromal tumors are predicted by different prognostic factors: a European Organisation for Research and Treatment of Cancer-Italian Sarcoma Group-Australasian Gastrointestinal Trials Group study. J Clin Oncol. 2005 Aug 20;23(24):5795-804. doi: 10.1200/JCO.2005.11.601. PMID 16110036
- [Background] Patyna S, Peng G. Distribution of sunitinib and its active metabolite in brain and spinal cord tissue following oral or intravenous administration in rodents and monkeys. European Journal of Cancer Suppl 4(12):21(Abstract 56), 2006.
- [Background] http://www.rxlist.com/cgi/generic/sutent
- [Background] http://www.pfizer/download/uspi_sutent.pdf
- [Background] http://ctep.cancer.gov/forms/CTCAEv3.pdf
- [Background] http://ctep.cancer.gov/guidelines/recist.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment goal was to enroll five participants; however, the study was terminated after only two participants had been enrolled as a result of slow recruitment and adverse events. Date of enrollment of the first participant was December 10, 2008, and the study was terminated on December 1, 2010.
Groups:
- Sunitinib Malate: Participants were expected to receive 9 months of sunitinib malate therapy administered in 6 cycles. Each cycle consisted of a daily oral dose of 50 mg sunitinib malate for 4 weeks followed by a 2-week rest period). Only one participant remained in the study for the Week 36 measures.
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 48.5 (4.95) [45 to 52]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Best Corrected Visual Acuity (BCVA) From Baseline to Week 36
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
Time Frame: Baseline and 36 Weeks
Measure: Number; unit: ETDRS Letters
Arm/Group | Left Eye | Right Eye
Number analyzed (Participants) | 1 | 1
ETDRS Letters | 1 | -5

2. Secondary Outcome: Change in Retinal Thickness From Baseline to Week 36
Description: Retinal thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
Time Frame: Baseline and 36 Weeks
Measure: Number; unit: µm
Arm/Group | Left Eye | Right Eye
Number analyzed (Participants) | 1 | 1
µm | 116 | 1

3. Secondary Outcome: Reduction in Leakage Intensity as Measured by Fluorescein Angiography From Baseline to Week 36
Description: Number of participants with improvement in leakage intensity.
Time Frame: Baseline and 36 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 2
Participants | 1

4. Secondary Outcome: Visual Field Changes as Documented by Microperimetry From Baseline to Week 36
Time Frame: Baseline and 36 Weeks
Population: Microperimetry was not accurate for any participants due to fixation issues so no data was collected. As such, zero participants were analyzed for this outcome.
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 0

5. Secondary Outcome: Changes in Non-ocular VHL Lesion Status
Description: Count of participants with new non-ocular lesions present since baseline at any follow-up visit.
Time Frame: Duration of study
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 2
Participants
  Renal: New Lesions Since Baseline | 0
  Renal: No New Lesions Since Baseline | 1
  Renal: N/A - Lesions Present at Baseline | 1
  Pancreatic: New Lesions Since Baseline | 0
  Pancreatic: No New Lesions Since Baseline | 1
  Pancreatic: N/A - Lesions Present at Baseline | 1
  Central Nervous System Hemangioblastoma: New Lesions Since Baseline | 0
  Central Nervous System Hemangioblastoma: No New Lesions Since Baseline | 1
  Central Nervous System Hemangioblastoma: N/A - Lesions Present at Baseline | 1
  Pheochromocytomas: New Lesions Since Baseline | 0
  Pheochromocytomas: No New Lesions Since Baseline | 2
  Pheochromocytomas: N/A - Lesions Present at Baseline | 0
  Endolymphatic Sac Tumors: New Lesions Since Baseline | 0
  Endolymphatic Sac Tumors: No New Lesions Since Baseline | 2
  Endolymphatic Sac Tumors: N/A - Lesions Present at Baseline | 0

6. Secondary Outcome: Reduction in Leakage Area as Measured by Fluorescein Angiography at the Week 36 Visit
Description: Number of participants with improvement in leakage area.
Time Frame: Baseline and 36 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (3)
Dizziness (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 2 (3)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (2)
Chills (General disorders) | 2 (5)
Stomatitis (Gastrointestinal disorders) | 1 (2)
Temperature intolerance (General disorders) | 1 (1)
Nail disclouration (Skin and subcutaneous tissue disorders) | 1 (1)
Urine analysis abnormal (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood creatine phosphokinase decreased (Investigations) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (4)
Hypertension (Vascular disorders) | 1 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Tooth extraction (Surgical and medical procedures) | 1 (1)
Platelet count decreased (Investigations) | 2 (3)
Blood creatine decreased (Investigations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 1 (1)
Hair disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Glossodynia (Gastrointestinal disorders) | 1 (2)
Lip pain (Gastrointestinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin discomfort (Skin and subcutaneous tissue disorders) | 1 (2)
Sleep disorder (Psychiatric disorders) | 1 (1)
Oral discomfort (Gastrointestinal disorders) | 1 (1)
Glossitis (Gastrointestinal disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 2 (5)

LIMITATIONS AND CAVEATS:
Early termination of the trial resulted in a small number of participants being analyzed, and Microperimetry (MP-1) results were not accurate for either participant due to fixation issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No